CLINICAL TRIAL: NCT00765310
Title: The Role of R-alpha Lipoic Acid in Prevention of Atherosclerotic Vascular Disease
Brief Title: Lipoic Acid and Prevention of Heart Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oregon State University (Other)
Collaborators: Oregon Health and Science University (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Gerd Bobe, Principal Investigator, Linus Pauling Institute; Associate Professor, Department of Animal Sciences, Oregon State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AT002034-1 (7186); 5P01AT002034 (NIH)
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Atherosclerosis
Keywords: atherosclerosis; lipoic acid; thioctic acid; triglycerides; overweight; obesity; oxidative stress; inflammation
MeSH Terms: conditions — Atherosclerosis; Overweight; Obesity; Inflammation | interventions — Thioctic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lipoic Acid (Active Comparator): 600 mg R-alpha lipoic acid in morning on empty stomach (two 300 mg capsules)
  Interventions: Dietary Supplement: R-alpha lipoic acid
- Placebo (Placebo Comparator): Placebo two caps every morning on empty stomach
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: R-alpha lipoic acid — 600 mg in morning on empty stomach (two 300 mg capsules)
  Other Names: Thioctic acid, LA, lipoic acid
  Arms: Lipoic Acid
Dietary Supplement: Placebo — two capsules once daily in morning on empty stomach
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if a dietary supplement, R-alpha lipoic acid, is able to reduce risk factors such as body weight and high blood cholesterol levels in overweight or obese participants.

DETAILED DESCRIPTION:
The purpose of this study is to see if a dietary supplement, R-alpha lipoic acid, is able to reduce risk factors such as body weight and high blood cholesterol levels in overweight or obese participants.

Recruitment will be in the Portland, Oregon area.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60
* Overweight (BMI, 25.0-29.9 kg/m2) or obese (BMI, >30 kg/m2);
* Elevated plasma triglycerides (100-400 mg/dl);
* Weight stable for the last three months and at lifetime maximum;
* Exercise limited to 30 minutes 3 times a week or less;
* Hs-CRP level at baseline of ≤ 10 mg/L;
* Consuming ≤ 2 alcoholic drinks per day;

Exclusion criteria:

* Pregnant, breastfeeding, or planning to become pregnant before the end of the study.
* Having had acute medical conditions, such as hospitalizations or surgeries, at least three months prior to entry into the study
* Diagnosed as having diabetes (fasting glucose <125 mg/dl for entry), cardiovascular disease, congestive heart failure, angina, thyroid disorders, cancer, inflammatory disorders or renal, hepatic, or hematological abnormalities;
* Currently taking lipid-lowering drugs, anti-hypertensive drugs, insulin , or oral hypoglycemic agents, anti-inflammatory drugs, weight loss medications, or hormone replacement therapy;
* On an extreme diet and not maintaining a prudent diet;
* Currently taking vitamin or antioxidant supplements, including R-alpha lipoic acid, except standard multivitamin/mineral supplements containing not more than the Daily Value (DV) of the vitamins and minerals;
* Smoking within the last three months;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2009-04-01 (Actual); Primary Completion 2011-11-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Triglycerides | 12 weeks and 24 weeks

SECONDARY OUTCOMES:
Body weight and composition | 12 and 24 weeks
Markers of inflammation and oxidative stress | 12 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Bobe, PhD, Principal Investigator — Oregon State University; Jonathan Q Purnell, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Derived] Bobe G, Michels AJ, Zhang WJ, Purnell JQ, Woffendin C, Pereira C, Vita JA, Thomas NO, Traber MG, Frei B, Hagen TM. A Randomized Controlled Trial of Long-Term (R)-alpha-Lipoic Acid Supplementation Promotes Weight Loss in Overweight or Obese Adults without Altering Baseline Elevated Plasma Triglyceride Concentrations. J Nutr. 2020 Sep 1;150(9):2336-2345. doi: 10.1093/jn/nxaa203. PMID 32692358